CLINICAL TRIAL: NCT06876571
Title: Pivotal, Clinical Study for the Accuracy Evaluation of the IdentiClone Dx TRG Assay
Status: Not yet recruiting | Type: Observational
Sponsor: Invivoscribe, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IVS-109-001
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: T-Cell Lymphoproliferative Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Deidentified residual DNA samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- T-Cell Positive Lymphoproliferative Disorders: FFPE Samples for subjects with T-Cell Positive Lymphoproliferative Disorders
  Interventions: Diagnostic Test: IdentiClone Dx TRG Assay
- FFPE Samples for subjects Negative for T-Cell Lymphoproliferative Disorders: FFPE Samples for subjects Negative for T-Cell Lymphoproliferative Disorders
  Interventions: Diagnostic Test: IdentiClone Dx TRG Assay

INTERVENTIONS:
Diagnostic Test: IdentiClone Dx TRG Assay — The IdentiClone Dx TRG Assay ("Assay") is an in vitro diagnostic product intended for qualitative capillary electrophoresis based-detection of clonality in T-cell receptor gamma chain (TRG) gene rearrangements in Formalin-Fixed Paraffin-Embedded (FFPE) specimens as an adjunctive method for the diagnosis of T-cell lymphoproliferative disease. This qualitative, non-automated Assay is for use on the ABI 3500xL Dx and ABI 3500xL Genetic Analyzers.
  Other Names: IdentiClone Dx IGH (IC IGH Dx) Assay

SUMMARY:
This protocol describes the pivotal accuracy study for the IdentiClone Dx TRG Assay. The intent of the accuracy study is to demonstrate agreement between the results of the IC TRG Dx Assay and a predicate devise or assay on retrospective and residual de-identified DNA extracted from FFPE (Formalin Fixed Paraffin Embedded) samples from individuals with suspected T-Cell Lymphoproliferations. The predicate device will be the LymphoTrack Dx TRG (FR1/FR2/FR3) Assays - MiSeq (LT Dx TRG-CE-IVD), which is a CE-IVD assay with a similar intended use as the IC TRG Assay on the same sample type.

ELIGIBILITY:
Inclusion Criteria:

1. De-identified, residual FFPE specimens with a minimum of 8 curls
2. Subject Age ≥ 18
3. For suspected clonal positive specimens, FFPE specimens of subjects diagnosed (at the time the specimen was drawn) with T-cell Lymphoproliferative disease with at least one of the following:

   1. ICD10 Codes: C84, C85.8, C85.9, C86.1, C86.2, C86.3, C86.5, 86.6, C91.5, C91.6, C91.0, C91.z, C91.9, C94, C95, C96, or other T-cell lymphoma diagnosis
   2. b. T-cell lymphoproliferative disease diagnosis per collection site procedure (e.g., SNOMED)
   3. Mycosis fungoides or Sézary syndrome sample are acceptable
4. For suspected clonal negative specimens, FFPE specimens of subjects suspected of T-cell lymphoproliferative disease but diagnosed negative for T-cell lymphoproliferative disease. Up to 20% of the negative specimens may be from normal tissue or tissue diagnosed with diseases other than T-cell lymphoproliferative disease

Exclusion Criteria:

1.FFPE specimens that were fixed using formalin substitute (ethanol, methanol, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples from subjects with diagnosed T-Cell Lymphoproliferative disorders or suspected of T-Cell Lymphoproliferative disorders with negative T-Cell Clonality Testing results
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-06-02 (Estimated); Primary Completion 2025-11-06 (Estimated); Study Completion 2025-12-06 (Estimated)

PRIMARY OUTCOMES:
% Agreement | Through Study Completion at one year
  Agreement between the results of the Invivoscribe IdentiClone Dx TRG Assay and the LymphoTrack Dx TRG (FR1/FR2/FR3) Assays - MiSeq by assessing the positive and negative percent agreement between the two assays.

CONTACTS AND LOCATIONS:
Locations (3):
- Invivoscribe, Inc., San Diego, California, United States
- LabPMM GmbH, Hallbergmoos, Germany
- LabPMM GK, Kawasaki-shi, Kanagawa, Japan

IPD SHARING:
Plan to Share IPD: No